CLINICAL TRIAL: NCT01589562
Title: A Randomized, Open Label, Single Dose, Cross-over, Phase I Trial to Investigate Safety and Pharmacokinetics of DW-ES(B) and Megace® Under Fed Conditions in Healthy Male Volunteers
Brief Title: Phase 1 Study of Daewon-ES(B) & Megace in Healthy Male Volunteers Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DW-ES 1201
Record Dates: First submitted 2012-04-24; First posted 2012-05-02 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
MeSH Terms: interventions — Megestrol Acetate; Megestrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Megace 800mg/20ml (Active Comparator): Fed condition
  Interventions: Drug: Megace 800mg/20ml
- DW-ES(B) 625mg/5ml (Experimental): Fed condition
  Interventions: Drug: DW-ES(B) 625mg/5ml

INTERVENTIONS:
Drug: Megace 800mg/20ml — Megestrol acetate 800mg/20ml, Suspension, Single dose
  Other Names: Megestrol; Megestrol Acetate
  Arms: Megace 800mg/20ml
Drug: DW-ES(B) 625mg/5ml — Megestrol acetate 625mg/5ml, Nano suspension, Single dose
  Other Names: Megestrol; Megestrol Acetate
  Arms: DW-ES(B) 625mg/5ml

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics of Daewon DW-ES(B) 625mg/5ml and Megace 800mg/20ml in healthy male volunteers under fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 40 years at screening.
* No significant congenital/chronic disease. No symptoms in physical examination.
* Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.
* History of taking megestrol

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
AUC of Megace 800mg/20mL | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120 hours post-dose
AUC of DW-ES(B) 625mg/5mL | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120 hours post-dose
Cmax of Megace 800mg/20mL | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120 hours post-dose
Cmax of DW-ES(B) 625mg/5mL | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 96, 120 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea